

# Sustained Treatment of Paroxysmal Atrial Fibrillation Post-Approval Study (STOP AF PAS)

Statistical Analysis Plan

Version 2 15 June 2017

Project Statistician: Christopher Anderson



# TABLE OF CONTENTS

| 1 | PURPOSE | 3 |
|---|------------------------------------------------------------------|----|
| 2 | RATIONALE FOR STUDYDESIGN | 3 |
| | 2.1 Stud y Purpose | |
| | 2.2 Stud y Scope | |
| | 2.3 System Description | |
| | 2.4 Data Collection | |
| 3 | DESCRIPTION OF ANALYSIS | 6 |
| | 3.1 General Summaries | 6 |
| | 3.1.1 Analysis Sets | |
| | 3.1.2 Use of Adjudicated Data | |
| | 3.1.3 Description of Baseline Variables | |
| | 3.1.4 Special Considerations | |
| | 3.1.5 Reports for which this Statistical Analysis Plan applies | |
| | 3.2 Primary Objectives | |
| | 3.2.1 Primary Objective #1 (Primary Effectiveness Objective) | |
| | 3.2.2 Primary Objective #2 (Primary Safety Objective) | 10 |
| | 3.3 Secondary Objectives | |
| | 3.3.1 Secondary Objective #1 (Effectiveness Objective) | |
| | 3.3.2 Secondary Objective #2 (Major Atrial Fibrillation Events.) | |
| | 3.3.3 Secondary Objective #3 (Long Term Safety Outcomes) | |
| | 3.3.4 Secondary Objective #4 (Cryoablation) | |
| | 3.3.5 Secondary Objective #5 (Procedure and Fluoroscopy Time) | |
| | 3.3.6 Secondar y Objective #6 (Adverse Events/Other) | 17 |
| | 3.4 Additional Analyses | |
| | 3.4.1 Additional Analysis Objective #1 | 17 |
| 4 | APPENDIX | |
| | 4.1 Overall Sample Sze | |
| | 4.2 General Statistical Considerations | |
| | 4.3 Interim Subject Safety Monitoring | |
| | 4.4 Sensitivity Analyses | |
| | 4.5 Acronyms | |
| | 4.6 References | 20 |
| _ | VEDGON HISTORY | 20 |

#### 1 PURPOSE

This Statistical Analysis Plan (SAP) has been designed to document the rationale for the study design, and the planned analyses that will be included in study reports.

## 2 RATIONALE FOR STUDYDESIGN

# 2.1 Study Purpose

The pivotal trial(STOP-AF) of the Arctic Front® Cardiac Cryoablation Atheter System with the adjunctive use of the Freezor® MAX Cardiac Cryoablation Catheter to electrically isolate pulmonary veins (PV) in patients with paroxysmal atrial fibrillation (PAF), compared to a randomized drug control grouphas been performed and a final report submitted to the FDA resulting inproduct approval December 2010. A Continued Access Protocol trial (CAPAF) was also conducted to allow collection of additional safety data following modifications implemented into the Arctic Front® Cathet and Cryoablation System. As part of the continued clinical development of the Arctic Front® rdiac Cryoablation Catheter System, this PostApproval Study (PAS) is being conducted to provide long-term safety and effectiveness monitoring/data per the Pe-Market Approval order (P100010) by the Food and Drug Administration (FDA).

This PAS is a prospective multicenter, non-randomized, single arm, controlled, unblinded clinical study of up to 400 enrolled subjects with PAF who have failed one or more Atal Fibrillation Drugs (AFDs). All study subjects will be receiving cryoablation with tstudy devices and, optionally (post-procedure), an Atrial Fibrillation Drug.

# 2.2 Study Scope

The study is expected to enroll subjects overan 18 - 24 month period with post procedural follow-up consisting of clinic visits a8, 6 and 12 months and 2 and 3 years. There was a CIP change in June of 2016 that reduced the followup time of this study from 5 years to 3 years. Prior to sites' activation of version 6 of the CHome subjects may also have been seen at 4 year or 5 year visits. This data will be included in the summary f safety outcomes.

Since the primary endpoint of the study is assessed at 3 years, the power of the study is not affected by this change.

More than 30 investigational sites in the United Statesand Canada have participated in this investigation. The Principal Investigator is Dr.Bradley Knight at Northwestern Memorial Hospital in Chicago, Illinois.

# 2.3 System Description

The investigational devices to be used in this trial are formally defined in the STOP AF PAS CIP version 6 (30JUN2016) Section 3. These devices include:

Arctic Front® Cardiac CyoAblation System, consisting of:

- Arctic Front® Cardiac CyoAblation CatheterOR
- Arctic Front Advance™ Cardiac CryoAblation Catheter
- Manual Retraction Kit
- The Freezor® MAX Cardiac CryoAblation Catheter
- Medtronic CryoCath CryoConsole

## 2.4 Data Collection

Clinical data are required to be collected at baseline/enrollment, procedure, post procedure, discharge, month (3, 6) followup, and year (1, 2, 3) followup. If a subject exits early, then a termination visit will also be conducted. The overall study design is summarized in Figure 1.



Figure 1: STOP AF PAS Overall Study Design

This SAP is based on Version6 of the STOP AF PAS Clinical Investigation Plan (30JUN2016).

#### 3 DESCRIPTION OF ANALYSIS

#### 3.1 General Summaries

#### 3.1.1 Analysis Sets

**Enrolled Set:** any subjects who have a signed informed consent.

Intent-To-Treat Set (ITT): any enrolled subjects who meet all inclusionand exclusion criteria.

mITT (modified intent-to-treat) Set: any subjects within the ITT setwith an Arctic Front® Cardiac CryoAblation Catheter System inserted into the vasculature for the purpose of this study.

All Treated Set: any subjects who have signed informed consent and have an Arctic Front® Cardiac CryoAblation Catheter Setem inserted into the vasculature.

## 3.1.2 Use of Adjudicated Data

For endpoint events that are to be adjudicated, only data fully adjudicated by the Adverse Event Adjudication Committee (AEAC) will be used in summaries and analyses AEAC determination of Chronic Treatment Failure (CTF), Cryoablation Procedure Events (CPE), and Major Atrial Fibrillation Event (MAFE), and their respective onset dates, are what the endpoint analyses utilizing these events will be based on. For adverse events (AE) reporting, AEAC determination of seriousness, and relatedness status will be used. Note that for data freezes and analyses before the final report it may not be possible for all data used to be adjudicated.

#### 3.1.3 Description of Baseline Variables

The following baseline disposition and procedural parameters reported on the case report forms (CRF) will be analyzed descriptively.

- The baseline and demographic characteristics, including but notimited to age, gender, race, height, weight, body mass indexrelevant medical history, arrhythmic symptoms, comorbid conditions, cardiovascular medical history, and concomitant medications. The baseline demographic tables will be reportetor both the ntent-To-Treat (ITT) Set and Modified Intent-To-Treat (mITT) Set.
- Subject disposition (analysis set allocation, discontinued along with primary reason for discontinuation, etc.) will be summarized using frequency and percent. A summary of subjects enrolled by site will be provided.

 A summary of Cryoablation procedure information including Oyoablation parameters (number, duration, average temperature, etc.),cryocatheter insertion time, PV ablation time, and total fluoroscopy time will be summarized basen the modified intent-to-treat (mITT) set

Tables and descriptive statistics will be used to summarize subject data with respect to these variables. For quantitative variables, number of nemissing observations, mean, median, minimum, maximum and standard deviation will be calculated. For qualitative variables, percentages and counts will be calculated.

#### 3.1.4 Special Considerations

# 3.1.4.1 Pooling of Study Centers for Analysis

A study center is defined as a treatment administration site or group of treatment administrative sites under the control and supervision of the same Principal Investigator. Each study center will be limited to enrolling no more than 50 subjects into the mITT set. Each center will be encouraged to enroll at least 10 subjects into the mITT. Set will prevent any single center from contributing a significant proportion of the subjects to the study. While every effort will be made to acquire similar enrollment from all participating centers, it is likely that some centers may enroll small routing of subjects. Therefore (for assessment of heterogeneity only) the centers that contribute five or fewer subjects to the mITT dataset will be pooled into a single 'super center'. The participating centers with more than five subjects in the mITT datastewill be reported individually.

Assessments of heterogeneity will be performed for the primary fectiveness and safety objectives across the investigational study centers. Analys of heterogeneity in primary endpoints will be conducted only in their fial report.

The level of heterogeneity of prepecified primary endpoints will be conducted using a random-effects meta-analytic approach. The R statistical software platform will be used to evaluate whether sites exhibit significant heterogeneity in entrates. If a Cochran's Gest for heterogeneity shows p<0.15, it will be taken as evidence of heterogeneity between sites. Evidence of betweensite heterogeneity will not preclude pooling data; rather, it may result in further investigation into the souces of the apparent differences in event rates between sites. In addition, a graphical display (such as a forest plot) of the proportions of primary effectiveness events and primarysafety events along with 95% confidence intervals for each center may beonstructed.

#### 3.1.4.2 Missing Data

The impact of missing data on the analysis of primary effectiveness and safety objectives is expected to be small sincehe Kaplan-Meier method will be performed for the primary objectives. For subjects who are lost to followp, the time to event will be censored at the last contact date.

Analysis will be based on available casesThe reasons for study withdrawal will be documented. There are no plans for imputation of any missing dataHowever, we will compare differences in baseline characteristics between subjects with complete data and subjects with early exit. Also, if the primarybjectives are met (p < 0.05) at 3 years, with >

5 subjects exiting prior to the-spear follow-up, a tipping point analysis will be conducted to assess sensitivity to missing data. Missing data is defined here as subjects with less than 3 years of follow-up.

Data will be sorted by ascending event times, and subjects who are censored prior to the 3-year visit are assigned an event time equal to a feet of last contact-index ablation date). Then, for each observation:

- 1) If the observation is censored, set time = time + 1 and event = 1.
- 2) Apply the logrank test (specified in section 3.2.1 or 3.2.2 for effica@and safety, respectively) to find the new twosided p-value and 95% loglog confidence interval.

The first observation where the confidence interval includes the performance goal (and the corresponding p-value  $\geq 0.05$ ) is the tipping point for the primary safety assisty For either primary endpoint, if fewer than 5 subjects have missing data, a worsets analysis will be done instead of a tipping point analysis. This analysis will be performed in the mITT datas et.

## 3.1.5 Reports for which this Statistical Malysis Plan applies

This analysis plan applies to the study final report, attore analysis results may be reported in study-related publications and interim progress reports Statistical analysis for study-related publications will not be limited to those defined in this plan.

# 3.2 Primary Objectives

The study will be considered a success if both primare ffectiveness and safety objectives are met at onesided 0.025 level of significance in the final nalysis. The analysis will be conducted using all mITT subjects.

#### 3.2.1 Primary Objective #1 (PrimaryEffectiveness Objective)

The primary effectiveness endpoint is the rate of subjects free of chronic treatmemiture (CTF) at 36 Months.

#### 3.2.1.1 Hypothesis

The following hypothesis will be tested in a onesided test at the 0.025 significance level.

Ho: Pe ≤ 45%

Ha: Pe > 45%

where Pe is the probability of freedom from CTF at 36 months and 4% is the prespecified performance goal based on theower bound of 95% CI for the primare ffectiveness rate in the STOP AF study.

#### 3.2.1.2 Endpoint Definition

Chronic Treatment Failure is defined as:

 Documented atrial fibrillation lasting longer than 30 seconds (outside the 90 day blanking period) OR  Intervention for atrial fibrillation (except for repeat cryoablation during the 90 day blanking period)

Intervention for atrial ibrillation is defined as: An invasive procedure intended for the definitive treatment of AF, including any ablation of the PVs or atrial triggers (other than protocol-specified ablation), interruption of AV nodal function, procedures to alter left atrial conduction or function such as the Maze procedure, or the implantation of an atrial pacemaker or atrial defibrillator; whether approved by relevant regulatory authorities or not for such indications; excluding electrical or pharmacologic cardioversion of rehythmias and excluding procedures solely directed at the treatment of atrial flutter or atrial tachycardias. A reablation permitted under Section 5.12 ofthe protocol is not an AF intervention.

#### 3.2.1.3 Analysis Methods

#### A. Statistical Methodology

The Kaplan-Meier method will be used to estimate the probability of chronic treatment success at 36 months followup. The standard error will be approximated using Greenwood's formula. A two-sided 95% log-log confidence interval for the probability will be constructed. The Kaplan-Meier estimate and its 95% log-log confidence interval will be constructed from the day of protocol specified ablation procedure D(ay 0) through the end of follow-up. For subjects with a treatment failure, the days of follow will be computed as the days from Day 0 to the failure date. For subjects without failure events, days of follow up will be computed as the days from Day 0 through the last follow-up. For subjects who are lost to follow-up, the last contact date will be used at follow-up date.

The survival curve will be presented through 36 months. Note that the phrases 'at 36 months' and 'through 36 months as used throughout includes events from the 3 year visit, even when it occurs more than  $3 \times 365 = 1,095$  days on the start date. The 36 month visit may occur after 1,095 days since the visit window runs until 30 daypast day 1,095. Rhythm monitoring that was initiated at the 36 month visit will be included in the analysis of the 36 month endpoint provided that the date of the documentation is no later than 30 day after the 36 month visit. Therefore, depending on the date of the 3 year visit, it is possible to include documentation as late as day 1,155. Not including such events after day 1,095 could underestim ate the proportion at 3 years due to 36 month visits that occur after 1,095 days. This potential bias is addressed in the statistical analysis by considering the date of recurrence to be exactly 36 months from the study ablation procedure so that these reflective will be counted as CTF in the 36 nonth Kaplan-Meier analysis.

## B Determination of Subject s/Data for Analysis

The analysis willbe conducted using the modified intent-to-treat (mITT) set.

#### 3.2.1.4 Sample Size Methods and Assumptions

Sam ple size was estimated using SAS v9.2 Proc Power. The sample size wasalculated under an asymptotic z-test for a single binomial proportion with continuity adjustment under the following assumptions:

Power = 90%, Sgnificance level = 0.025 (one ided), Assumed underlyin g effectiveness rate = 55%, Performance goal = 45%.

Long-term (> 12 months) effectiveness of pulmonary vein isolation for ttreatment of atrial fibrillation (AF) ranges from 4470%, with 40% reported as theninimum goal by physicians¹. Shah et al reported that the annual rate of atriaflbrillation recurrence after one year was 8.8% and ₹ou et al reported a similaannual rate of 7%³³. Based on the STOP AF results and assuming an annual rateof atrial fibrillation recurrence of -₹9%, the estimated effectiveness rate at 36months would be approximately 55%. Theperformance goal of 45% wasdetermined from the lower bound of 95% CI for the primare/ffectiveness rate in STOP AF study.

Figure 2 presents the sample size at different primary ffectiveness rates under the assumptions outlined above.



Figure 2. Sample Size vs. Primary Effectiveness Rate

If the underlying effectiveness rate is assumed 55%, a total of 270 evaluable subjects will be required to provide 90% power to meet this effectiveness objective.

#### 3.2.2 Primary Objective #2 (Primary Safety Objective)

The primary safety endpoint is the rate of subjects experiencing one or m@eyoablation Procedure Events (CPE) through 12 months.

#### 3.2.2.1 Hypothesis

If the upper bound of the confidence interval for CPE rate at 12 months is less than the performance goal of 14.8%, we can conclude the primary safety objective is met.

The following hypothesis will be tested in a orseided test at the 0.025 significance level.:

Ho: Ps≥ 14.8% Ha: Ps < 14.8%

where Ps is the probability of subjects with one or more CPhed at 4.8% is the pre specified performance goal based on the upper bound of 95% CI for the primærayfety rate in the STOP AF study.

## 3.2.2.2 Endpoint Definition

A CPE is a devicerelated or procedure-related serious adverse event (SAE) with onset between the timeof the subject's entry into the procedure room for the studyspecified cryoablation procedure (Day 0) through the indicated onset intervals as set out in the following Table 1:

Table 1: Cryoablation Procedure Events

| Cryoablation Procedure Events (CPIs) | Onset Interval |
|------------------------------------------|-------------------|
| Access site complications requiring: | Through 7 days |
| Transfusion of 3 or more units or | |
| Surgical intervention or | |
| Permanent loss or functionalimpairment | |
| Cardiac damage (including MI) except for | Through 7 days |
| Pulmonary vein stenosis* | Through 12-months |
| Atrio-esophogeal fistula | Through 12-months |
| Embolic complications (including stroke) | Through 7 days |
| Arrhythmias | Through 7 days |
| Persistent phrenic nerve palsty* | Through 12-months |
| Death | Through 7 days |

<sup>\*</sup> CPE will be assessed at the completion of the follow visit, as determined by CT/MRI Core Lab.

- Pulmonary vein stenosis is defined as > 75% reaction in the baselinearea after 6-month follow-up.
- Phrenic nerve palsy (alternatively, Phrenic Nerve Injury or PNI)s defined as abnormal diaphragm excursion as demonstrated during the postcryoablation procedure fluoroscopy. PNI events are considered persistent if they are unresolved at 12 months. CPEs exclude
  - 1. Adverse events that are normal and expected concomitants of catheterization and diagnostic and ablation electrophysiology (EP) procedures, such as induced arrhythmia and groin ecchymosis, bu only IF that AE resolves completely AND involves only routineresponses such as medication, fluids, compression, temporary pacing, or cardioversion.
  - 2. Atrial fibrillation or atrial flutter occurring during postirocedural hospitalization.
- CPEs will be accrued for Retreated Subjects for the comparable 7 day period following a repeat cryoablation.

<sup>\*\*</sup> CPE will be assessed at the completion of the foll-top as determined by chest X-ray (insp/exp)

## 3.2.2.3 Analysis Methods

#### A. Statistical Methodology

The Kaplan-Meier method will be used to estimate the probability of a subject experiencing one of more CPE at 12 months followup. The standard error will be approximated using Greenwood's formula. A two-sided 95% log-log confidence interval for the probability will be constructed. The Kaplan-Meier estimate and its 95% log-log confidence interval will be constructed from the day of study specified cryoablation procedure Day 0) through the end of follow-up. For subjects with safety events, the days of follow-p will be computed as the days from Day 0 to the onset date of the first safety event. For subject without safety events, days of follow-p will be computed as the days from Day 0 through the last follow-up. For subjects who are lost to follow-p, the last contact date will be used as the last follow-up date.

The 12 month visit may occur after 36days since the visit window runs until 30 days past day 365. Not including eventsthat result from assessment at a 12month visit, but after day 365 could underestimate the proportion at 1 year due to 12 month visits that occur after 365 days. This potetial bias is addressed in the statistical analysis by considering the date of recurrence to be exactly 12 month (365 days) from the study ablation procedure so that these events will be counted a PE in the 12-month Kaplan-Meier analysis.

#### B Determination of Subject s/Data for Analysis

The analysis willbe conducted using the modified intent-to-treat (mITT) set.

#### 3.2.2.4 Sample Size Methods and Assumptions

Sam ple size was estimated using SAS v9.2 Proc Power. The sample size was calculated under an asymptotic z test for a single binomial proportion with a continuity adjustment under the following assumptions:

Power = 90%, Significance level = 0.025 (oneided), Assumed underlying primary safety event rate = 6%, Performance goal = 14.8%.

The performance goal of 14.8% is selected ased on the same assumption defined in version 1.7 of the STOP AF Clinical Investigation plan (January ,152008): "Based on a review of SEEDs for similar types of ablation trials, the expected rate for CPEs in a well-monitored trial of left atrial RF ablation for AF was estimated to be 10% (corresponding to a CPEfree rate of 90%). If 16 of 160 subjects were observed to have at least one CPEs then the resulting onesided 95% upper confidence bound would be 14.8%."; where SEED is an abbreviation for Summary of Safety and Effectiveness Data.

Figure 3 presents the sample size at different primarsyafety event rates under the assumptions outlined above.



Figure 3. Sample Size vs. Primary Safety Event Rate

If the underlying safety event rate is assumed 6%, a total of 14ed valuable/mITT subjects will be required to provide 90% power to meet this safety objective.

# 3.3 Secondary Objectives

All secondary analyses will be exploratory and no formal hypotheses tested.

## 3.3.1 Secondary Objective #1 (Effectiveness Objective)

The probability of subjects free of chronic treatment failure at the 4nd 2 yearfollow-up visits will be estimated.

#### 3.3.1.1 Hypothesis

There is no hypothesis.

## 3.3.1.2 Endpoint Definition

Chronic treatment failure is defined in Primary Objective #1, section 3.2.1.2. Subjects free of chronic treatment failure are those that do not meet that definition.

#### 3.3.1.3 Analysis Methods

#### A. Statistical Methodology

The Kaplan-Meier method will be used to estimate the probability of chronic treatment success at 1 and 2 yearfollow-ups. The standard error will be approximated using Greenwood's formula. Two-sided 95% log-log confidence intervals for the probability will be constructed for each of the four followups. The Kaplan-Meier estimates and their 95% log-log confidence intervals will be constructed from the day of protocol specified ablation procedure (Day 0) through the end of followup. For subjects with a treatment failure, the days of follow-up will be computed as the day from Day 0 to the failure date. For subjects without failure events, days of follow-up will be computed as the days from Day through the last follow-up. For subjects who are lost to follow-up, the last contact date will be used as the last follow-up date.

## B Determination of Subject s/Data for Analysis

The estimations will be conducted using the modified intentto-treat (mITT) set.

# 3.3.2 Secondary Objective #2(Major Atrial Fibrillation Events)

The probability of subjects free of Major Atrial Fibrillation Events (MAFE) at the 1an2d, 3 year follow-up visits will be etimated.

# 3.3.2.1 Hypothesis

There is no hypothesis.

#### 3.3.2.2 Endpoint Definition

Major Atrial Fibrillation Event (MAFE): A MAFE is a serious adverse event (SAE) which has not been categorized as a CPE as set out in the following table:

Table 2: Major Arial Fibrillation Events

| Table 2. Major Alai I Ibililation Events |
|------------------------------------------------|
| Major Atrial Fibrillation Events (MAFEs): |
| Cardiovascular deaths |
| Hospitalizations for (primary reason): |
| AF recurrence or ablation |
| Atrial flutter ablation (excluding Type I) |
| Systemic embolization (not stroke) |
| Congestive heart failure |
| Hemorrhagic event (not stroke) |
| Antiarrhythmic drug: initiation, adjustment or |
| complication |
| Myocardial infarction (MI) |
| Stroke |

## 3.3.2.3 Analysis Methods

#### A. Statistical Methodology

The Kaplan-Meier method will beused to estimate theprobability of a subjectbeing free of MAFE at 1, 2, and 3 yearfollow-ups. The standard error will be approximate using Greenwood's formula. Two-sided 95% log-log confidence intervals for the probability will be constructed for each of the five followups. The Kaplan-Meier estimates and their95% log-log confidence intervals will be constructed from the day of study specified cryoablation procedure (Day 0) through the end of each follow-up. For subjects with MAFE, time until an event will be computed as the number of days from Day 0 to the onset date of the first MAFE. For subjects withouta MAFE, the number of days at-risk will be computed as the days from Day 0 through the lastime they had an opportunity to report a MAF, which includes scheduled study follow-up visits and their associated testing plus the termination visit, if done For subjects who are lost to follow-up", time from Day 0 untilast contact date will be used as the number of days at risk.

## B Determination of Subject s/Data for Analysis

The estimations will be conducted using the modified intentto-treat (mITT) set.

#### 3.3.3 Secondary Objective #3(Long Term Safety Outcomes)

Device and procedure related events, serious adverse events(SAE), and other safety categories will be collected through the 3 year follow-up and reported descriptively.

#### 3.3.3.1 Hypothesis

There is no hypothesis.

#### 3.3.3.2 Endpoint Definition

Device and procedure related events, and SAEs are defined in section 7.2.1 of IP version 6.

#### 3.3.3.3 Analysis Methods

#### A. Statistical Methodology

For each event, the total number of events, the number of subjects with at least one event, and the percentage of subjects with at least one event will be reported. Totals and sub totals will be reported in the same manner. Il of these events will be categorized using the MedDRA or similar system, tabulated and listed in decreasing frequency order.

#### B Determination of Subject s/Data for Analysis

The population(s) used for descriptive summarization will be the mITT set.

#### 3.3.4 Secondary Objective #4(Cryoablation)

Cryoablation procedure parameters will be summarized

#### 3.3.4.1 Hypothesis

There is no hypothesis.

#### 3.3.4.2 Endpoint Definition

- Cryoablation procedure parameters such as total number of coyablation attempts, mean number of cryoablation attempts per attempted subject and number of successful cryoablations per subject will be summarized using descriptive statistics.
- Cryoablation temperature and ablation procedure time (duration) will be summarized using descriptive statistics.

#### 3.3.4.3 Analysis Methods

# A. Statistical Methodology

Tables and descriptive statistics will be used to summarize subject data with respect to these variables. For quantitative variables, number of nemissing observations, mean, median, minimum, maximum and standard deviation will be calculated. For qualitative variables, percentages and counts will be calculated. Summaries for index ablation and retreatment procedures will be reported separately. Categories of 'other' will be reported in associated listings.

For the final report, most of the statistics reported will describe subjected phenomena, requiring aggregation (for example, by taking the average, minimum or maximum) when measurements such as cryoablation temperature are recorded in the data at the or application level.

#### B Determination of Subject s/Data for Analysis

The population used for descriptive statistics will be the mITT set.

#### 3.3.5 Secondary Objective #5(Procedure and Fluoroscopy Time)

Total procedure time and total fluoroscopy time willbe summarized.

#### 3.3.5.1 Hypothesis

There is no hypothesis.

#### 3.3.5.2 Endpoint Definition

- Total procedure time defined as the period from puncture of the skin performed to obtain venous access for catheter placement to final ECG (electrocardiogram) at end of procedure will be analyzed using descriptive statistics.
- Total fluoroscopy time will be analyzed using descriptive statistics.

#### 3.3.5.3 Analysis Methods

#### A. Statistical Methodology

Tables and descriptive statistics will be used to summarize subject data with spect to these variables. The number of normissing observations, mean, median, minimum, maximum and standard deviation will be calculated. Summaries for index ablation and re treatment procedures will be reported separately.

## B Determination of Subjects/Data for Analysis

The population used for descriptive statistics will be the mITT set.

## 3.3.6 Secondary Objective #6 (Averse Events/Other)

All adverse events will be summarized.

## 3.3.6.1 Hypothesis

There is no hypothesis.

#### 3.3.6.2 Endpoint Definition

All adverse everts that occur during the study will be captured on the CRFs.

#### 3.3.6.3 Analysis Methods

#### A. Statistical Methodology

All adverse events will be summarized by presenting the number of events, the number and percentage of subjects having any AE, having anEAin each body system, and having each individual AE. Any other information collected (e.g., seriousness, severity or relatedness to device/procedure) will be presented as appropriate.

#### B Determination of Subject s/Data for Analysis

The population used for descriptive statistics will be the enrolled set. Summaries will be presented for both the IntentTo-Treat (ITT) Set and Modified IntentTo-Treat (mITT) Set

## 3.4 Additional Analyses

#### 3.4.1 Additional Analysis Objective #1

Though not defined as an objective in the CIP, a posthoc analysis on SF-12 Health Survey scores collected at baseline, 6 month, 12 month year, and 3 yearvisits will be included in the Final Report

#### 3.4.1.1 Hypothesis

There is noformal statistical hypothesis associated with this objective

#### 3.4.1.2 Endpoint Definition

There are two endpoints associated with this objective: the SF2 physical health component score and the SF-12 mental health component score.

## 3.4.1.3 Analysis Methods

## A. Statistical Methodology

The Medical Outcome Study Short Form-12 (SF-12) questionnaire will also be utilized for this objective. The SF-12 questionnaire is a health-related quality of life questionnaire to evaluate the subject's mental and physical performance. For each questionnaire, the physical and mental component scores were calculated using standard scoring algorithms that combine the survey item responses. Both the physical and mental component scores range from 0 to 100, where a 0 score indicates the lowest level of health measured by the scale and 100 indicates the highest level of health.

Summary statistics (e.g. mean, SD, 95% confidence intervals) and graphical methods will be used to describe SF-12 scores from baseline through36 months. For a subject's physical health score to be calculated at eitherntie point, all physical health dimension questions must be answered; likewise, for mental health scores to be calculated, all mental health questions must be answered. Analysis will be performed on all complete questionnaires from subjects in the mITT datast.

#### 4 APPENDIX

#### 4.1 Overall Sample Size

In order to adequately power for both the primars effectiveness and safety hypotheses, we require a sample size of 270 evaluable subjects to complete 36 months of follow We estimate that the attrition rate will be proximately 10% per year for the duration of the originally intended 5 year follow-up period. Therefore, the final sample size required to achieve 270 subjects followed for 36 months and account for attrition (i.e. 10% per year) is 370 mITT subjects with pocedure attempts. It is expected up to 400 subjects will need to be enrolled to ensure 370 mITT subjects with procedure attempts assuming a small number of subjects who are enrolled will not undergo a procedure.

#### 4.2 General Statistical Considerations

All analyses will be performed using SAS statistical software (SAS Institute Inc, Cary, NC). It is planned that the data from all centers that participate in this protocol will be combined for analysis. Descriptive statistics includes but is limited to number of on-missing observations, mean, standard deviation, median, minimum, and maximum for continuous



variables and count and percentage for categorical variables. Unless otherwise specified, the analysis will be performed using descriptive statistics.

# 4.3 Interim Subject Safety Monitoring

No formal interim analyses are planned. However, accumulating data for the safety endpoints may be analyzed at any time per regulatory agents request. Hypothesis statistical testing will not be conducted until the final analysis. No alpha adjustment will be applied in terms of the analysis of the final primagndpoint for all subjects.

Note that incidence rate estimates from analyses for the interim reports malgrave some upward bias since subjects that recently had a 36-month visit that occurred prior to precisely 36 months will not part of the risk settlenominator) at 36 months due to being censored at their last followup.

# 4.4 Sensitivity Analyses

In the rare instance where a subject who has y@Ablation Catheter System treated but does not meet all inclusion and exclusion, the subject will not be included in ITT and mITT set. If deemed necessary, analyses performed on the mITT analysis set may be repeated based on all treated analysis set to assess sensitivity to the inclusion criteria.

# 4.5 Acronyms

| AE | adverse event(s) |
|--------|----------------------------------------------|
| AEAC | Adverse Event Adjudication Committee |
| AF | atrial fibrillation |
| AFD | atrial fibrillation drug(s) |
| CI | confidence interval |
| CIP | Clinical Investigation Plan (protocol) |
| CPE | cryoablation procedure event(s) |
| CRF | case report form(s) |
| CT | computed tomography |
| CTF | chronic treatment failure |
| ECG | electrocardiogram |
| EP | electrophysiology |
| FDA | Food and Drug Administration |
| ITT | Intent to Treat population |
| MAFE | major atrial fibrillation even(ts) |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | myocardial infarction |
| mITT | Modified Intent to Treat population |
| MRI | magnetic resonance imaging |
| PAF | paroxysmal atrial fibrillation |
| PV | pulmonary vein(s) |
| RF | radio frequency |
| SAE | serious adverse event(s) |
| SAP | statistical analysis plan |
| SAS | Statistical Analysis Systems (software) |
| SSED | Summary of Safety and Effectiveness Data |

STOP-AF Previous pivotal trial

UADE unanticipated adverse device effect(s)

#### 4.6 References

<sup>1</sup> Katritsis D, Wood M, Giazitzoglou E, Shepard R, Kourlaba G, Ellenbogen K. Lonterm follow-up after radiofrequency catheter ablation for atrial fibrillation. Europace. 2008;10:419424.

<sup>2</sup> Shah A, Mittal S, Schrovsky T, Cotiga D, Arshad A, Maleki K, Pierce, Waterinberg J. Long-term outcome following successful pulmonary vein isolation: pattern and prediction of very late recurrence. J Caridiovasc Electrophysiol. 2008;19:661-667.

J Caridiovasc Electrophysiol. 2008;19:661-667.

Tzou W, Marchlinski F, Zado E, Lin D, Dixit S, Callans D, Cooper J, Bala R, Garcia F, Hutchins M, Riley M, Verdino R, Gerstenfeld E. Longerm outcome after successful catheter ablation of atrial fibrillation. Circ Arrhythm Electrophysiol. 2010;3:237242.

fibrillation. Circ Arrhythm Electrophysiol. 2010;3:237242.

<sup>4</sup> Ware J, Kosinki MKeller S, A 12-Item Short Form Health Survey: construction of scales ad preliminary tests of reliability and validityMed Care. 1996; 34(3):220233.

# 5 VERSION HISTORY

| Version | Summary of Changes | Author(s)/Title |
|---|---|---|
| 1.0 | Not Applicable, New Document | Jian Huang |
| 2.0 | <ul> <li>Replaced assessments scheduled to take place at 5 years to refet new 3 year timeline of the study replaced 5-year outcomes with equivalent 3year outcomes.</li> <li>Modified the statistical methods for center pooling to accommodate 20-30 sites (replaced chi square test with Cochran's Q).</li> <li>Specified details about conducting the tipping point analysis</li> <li>Removed language pertaining to describing subject screening</li> <li>Removed additional objectives 1 and 2, which centered around comparing results between this study and the STOP AF Pivotal study, and are now considered out of scope.</li> <li>Specified an additional analysis describing SF-12 scores at baseline, six months, and at year 1, 2, and 3</li> </ul> | Christopher Anderson |